CLINICAL TRIAL: NCT04804176
Title: Study on the Mode and Mechanism of Ultra-low Frequency Repetitive Transcranial Magnetic Stimulation for Sleep Disorders in Patients With Parkinson's Disease
Brief Title: Study on the Mode and Mechanism of Ultra-low Frequency rTMS for Sleep Disorders in Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, Professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULFRTMS-S
Record Dates: First submitted 2021-03-08; First posted 2021-03-18 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Repetitive Transcranial Magnetic Stimulation; Parkinson Disease; Sleep Disorder
Keywords: repetitive transcranial magnetic stimulation; Parkinson's disease; sleep disorder
MeSH Terms: conditions — Parkinson Disease; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: The study was divided into three groups, which were control group, group A and group B.Groups A and B received different treatment modalities on the same device.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 5-HT mode of Ultra-low frequency repetitive transcranial magnetic stimulation (Active Comparator): The study used 5-HT mode of Ultra-low frequency repetitive transcranial magnetic stimulation for 35 minutes once a day.Every 7 days is a cycle.The stimulus intensity was 400GS.
  Interventions: Device: Ultra-low frequency repetitive transcranial magnetic stimulation
- GABA mode of ultra-low frequency repetitive transcranial magnetic stimulation (Active Comparator): The study used GABA mode of ultra-low frequency repetitive transcranial magnetic stimulation for 35 minutes once a day.Every 7 days is a cycle.The stimulus intensity was 400GS
  Interventions: Device: Ultra-low frequency repetitive transcranial magnetic stimulation
- the control group (Sham Comparator): The instrument is not working, only in exhaust mode.
  Interventions: Device: Ultra-low frequency repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Ultra-low frequency repetitive transcranial magnetic stimulation — Two different modes of the instrument were used to treat patients in groups, to compare the efficacy.

SUMMARY:
The study by giving a sleep disorder Parkinson's disease patients with different patterns of ultra-low frequency transcranial magnetic stimulation or sham stimulation, scale for assessment of the patients were observed, hematology and imaging changes before and after therapy, clear ultra-low frequency transcranial magnetic stimulation for sleep disorder Parkinson's disease treatment, to explore the mechanism of action, compare the difference between different modes.

DETAILED DESCRIPTION:
Parkinson's disease is the second most common chronic neurodegenerative disease.At present, researchers focus not only on the motor symptoms of Parkinson's disease, but also on the non-motor symptoms of Parkinson's disease (including mood disorders, sleep disorders, cognitive decline, and autonomic nervous kinetic disorder, etc.).The principle of transcranial magnetic stimulation is based on the electromagnetic principle proposed by Faraday. When an electrifying coil is suspended over the scalp at a certain distance, the magnetic field generated by the coil current and the electric field generated by the magnetic field can reach the skull and directly or indirectly affect the synapses and neurons in the brain.The study by giving a sleep disorder Parkinson's disease patients with different patterns of ultra-low frequency transcranial magnetic stimulation or sham stimulation, scale for assessment of the patients were observed, hematology and imaging changes before and after therapy, clear ultra-low frequency transcranial magnetic stimulation for sleep disorder Parkinson's disease treatment, to explore the mechanism of action, compare the difference between different modes.

ELIGIBILITY:
Inclusion Criteria:

* in line with international Movement disorders association (the Movement Disorder Society, MDS) in 2015 the diagnosis of Parkinson's disease diagnosis standard and China standard (2016)
* can cooperate to complete rating scale, the sleep monitoring, imaging and blood test
* have a sleep disorder
* aged 18 to 70 years old
* agree to participate in this experiment, and have signed the informed consent

Exclusion Criteria:

* superposition of diagnosed with Parkinson's syndrome
* secondary diagnosed Parkinson's syndrome
* is equipped with heart pacemakers and other metal implants
* cannot achieve scale assessment
* has significant malignant diseases
* has a history of seizures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-04-20 (Estimated)

PRIMARY OUTCOMES:
change from length of sleep at one week | one week
  Sleep duration was monitored by polysomnography.It's measured in minutes.
change from ratio of stage 3 sleep in total sleep at one week | one week
  The proportion of phase 3 sleep in total sleep was monitored by polysomnography.It's in percentages.
change from limb movement of sleep at one week | one week
  The number of body movements during sleep was recorded by polysomnography.It's in units of times per night.
change from nocturnal arousal frequency at one week | one week
  The number of nocturnal awakenings was recorded by polysomnography.It's in units of times per night.
change from Pittsburgh sleep quality index scale at one week | 1 day before treatment、1 day after treatment、1 week after treatment、1 moth after treatment
  The scale was evaluated on the day before treatment and the day after treatment, which was based on scores.The total score of the scale ranges from 0 to 2L, and the higher the score, the worse the sleep quality.
Interleukin 6 | 1 day before treatment and 1 day after treatment
  It plays an important role in central nervous system diseases. In PD, the increase of IL-6 is the body's self-defense mechanism to protect neurons, and the change of IL-6 in peripheral blood can reflect the change of injury aggravation and recovery.It is also associated with psychiatric symptoms, and IL-6 is elevated in major depression.
change from the Epworth sleepiness scale at one week | one week
  The scale was evaluated on the day before treatment and the day after treatment, which was based on scores.The scale has an overall score range of 0 to 24, with higher scores indicating more severe sleepiness.
change from Parkinson's disease sleep scale at one week | one week
  The scale was evaluated on the day before treatment and the day after treatment, which was based on scores.The total score of the scale ranges from 0 to 150. The higher the score, the better the sleep.
change from movement disorders association - comprehensive rating scale of Parkinson's disease at one week | one week
  The scale was evaluated on the day before treatment and the day after treatment, which was based on scores.The total score of the scale ranged from 0 to 260, and the higher the score, the more severe the symptoms were.
change from Parkinson's disease quality of life scale one week | one week
  The scale was evaluated on the day before treatment and the day after treatment, which was based on scores.The total score of the scale ranges from 0 to 156, and the higher the score, the worse the quality of life.
change from Hamilton depression scale at one week | one week
  The scale was evaluated on the day before treatment and the day after treatment, which was based on scores.The total score of the scale ranged from 0 to 96, and the higher the score, the more severe the depression was.
change from Hamilton anxiety scale at one week | one week
  The scale was evaluated on the day before treatment and the day after treatment, which was based on scores.The total score of the scale ranges from 0 to 56, and the higher the score, the more serious the anxiety.
change from simple mental state scale at one week | one week
  The scale was evaluated on the day before treatment and the day after treatment, which was based on scores.The total score of the scale ranges from 0 to 30, and the lower the score, the more severe the cognitive impairment.
change from Montreal cognitive assessment scale at one week | one week
  The scale was evaluated on the day before treatment and the day after treatment, which was based on scores.The total score of the scale ranges from 0 to 30, and the lower the score, the more severe the cognitive impairment.
change from magnetic resonance imaging of the brain at one month | one month
  The ADC values of sleep-related brain tissues were measured by diffusion weighted magnetic resonance imaging of the brain.Compare the difference between the measured results on both sides of the same site and record the difference.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuhua Li, MD, Principal Investigator — Qianfoshan Hospital，The First Affiliated Hospital of Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No